CLINICAL TRIAL: NCT01942278
Title: CIDRZ 1229- Better Health Outcomes Through Mentoring and Assessment (BHOMA)
Brief Title: Better Health Outcomes Through Mentoring and Assessment (BHOMA)
Acronym: BHOMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: CIDRZ 1229
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-02

CONDITIONS: Patient Care
Keywords: Healthcare; Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Care is delivered according to baseline standard practice
- BHOMA (Experimental): Care is delivered according to the BHOMA intervention
  Interventions: Other: BHOMA

INTERVENTIONS:
Other: BHOMA — A complex health systems, clinical care, and community intervention to improve outcomes
  Arms: BHOMA

SUMMARY:
BHOMA Interventions

The purpose of this study is to assess the impact of the BHOMA intervention on health in 3 rural districts of Zambia.

DETAILED DESCRIPTION:
The BHOMA study includes systematic program implementation designed to contribute to generalizable knowledge and evaluation of this program. The program aims to improve primary health care through an integrated package of interventions, at both health facility and community level, centered on improving the patient -provider interface which is considered to be key to improving health outcomes. The primary objective of this research is to assess the impact of the BHOMA intervention on health in three rural districts of Zambia.

Objectives include: to understand the causal pathways of the BHOMA interventions by analyzing inputs, processes, outputs, and outcomes; to measure the cost of the BHOMA interventions; and to measure whether the health system has been strengthened by the BHOMA interventions. The endpoints of the study will be measured by a combination of facility surveys, facility health worker and community health worker interviews, quality assessments, qualitative studies and community surveys.

The study involves 7 stepped introduction of the programme in 48 facilities. A step typically involves initiation of a set of selected health facilities and the communities they serve. On average, 6 randomly selected sites are involved in a step. Facility workers are trained; community health workers, clinic support worker and traditional birth attendants are identified and trained through a month-long Ministry of Health (MOH) approved course. Equipment for data collection and electronic capture are set up, filing systems established and the study begins when the tools get implemented. Close supervision is provided for at least a month following initiation; there after regular supervisory visits are done by six quality improvement teams.

Clinic Intervention, implemented by the Centre for Infectious Disease Research in Zambia (CIDRZ) BHOMA program:

The clinic intervention consists of the following 5 components: 1) the implementation of clinical care forms and accompanying job aids, 2) resources, to includes equipment, supplies, staffing and infrastructure, 3) clinic implementation, which involves a quality improvement team working at the clinic to introduce the new patient flow system and to improve the skills of clinic staff, 4) the use of electronic information for performance assessment, which involves implementing an electronic data entry system within the clinics and 5) supportive mentoring, which will involve the Quality Improvement (QI) team reviewing patient charts for appropriate screening, diagnostics, treatment or follow-up, attending patient visits, identifying equipment or infrastructure issues, and reviewing clinic performance reports and updating the clinic's quality improvement strategy.

Community Intervention, implemented by the CIDRZ BHOMA program:

The community intervention aims to expand the availability of community-based health services and improve the quality of these services with the use of three groups:

Community Health Workers:

The investigators will engage one community health worker (CHW) per Neighborhood Health Committee to conduct patient follow-up and household assessments. The CHWs will use two forms - patient follow-up form and a household assessment form, and will be trained to assess which patients need referral to the clinic or hospital.

Traditional Birth Attendants:

The investigators will offer training for traditional birth attendants (TBAs) working near the implementation clinics. The training will review the goals of facility delivery and introduce a pregnancy referral form for TBAs. The investigators will encourage the TBA to help the patient arrive at the clinic, and provide incentives for the TBAs for clinic referrals. The investigators will also train the TBAs to follow up all pregnancies in the first month to assess the infant and teach the mother about when it is appropriate to bring the infant to the clinic. TBAs will complete infant follow-up forms.

Neighborhood Heath Committees (NHC):

These committees will complete a community health event register, during which they will capture information about serious sicknesses and deaths that are not recorded at the clinics. Each NHC will visit households and return their register to the clinic.

These activities will continue throughout the duration of the funded project.

ELIGIBILITY:
Inclusion Criteria:

Intervention Sites The intervention will involve all of the health facilities in the Chongwe, Kafue and Luangwa districts.

Exclusion Criteria Hospitals will be excluded from the intervention as they do not have discrete catchment populations. The intervention will be implemented by 6 teams each of which will use 1 facility as a pilot site to test out the intervention. The pilot sites will be excluded from the evaluation. Health facilities with catchment populations exclusively serving the armed forces will be excluded.

Inclusion Criteria

* All enumerated adults who are able to give written, informed consent. If an adult is illiterate they may be asked to give consent providing the information is read to them and it is established that they fully understand its contents and there is a witness available to witness the understanding of the information and the fingerprinting of the consent form.
* All adolescents 10-17 years and children 5 years or less who have a parent or responsible guardian who is able to give written, informed consent. If the parent or guardian is illiterate they may be asked to give consent providing the information is read to them and it is established that they fully understand its contents and there is a witness available to witness the understanding of the information and the fingerprinting of the consent form.

Exclusion Criteria

* Any adult who is unable to give informed consent due to mental or other disability
* Any adolescent or child who has no responsible parent or guardian
* Any household member who has been absent from the house for more than 72 hours

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 207517 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Age standardized mortality rates in those aged <60 years. | 4 years
  The sample size is based on a mortality rate for those aged<60 years of 20/1000 person years, each of 3 cross sectional surveys recruits 150 households of whom 6 members are aged <60 years, and births and deaths within the household in the last 12 months are ascertained. For a values of k between 0.2 and 0.3 there is at least 90% power to detect a 35% reduction in mortality, and for k=0.35 there is approximately 87% power.

SECONDARY OUTCOMES:
Mortality in those aged <5 years. | 4 years
  The sample size is based on a mortality rate for those aged<5 years of 35/1000 person years (equivalent to under-5 mortality of 168/1000), each of 3 cross sectional surveys recruits 150 households of whom 2 members are aged <5 years, and births and deaths within the household in the last 12 months are ascertained. For a values of k between 0.2 and 0.3 there is at least 90% power to detect a 35% reduction in mortality, and for k=0.35 there is approximately 84% power.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Stringer, MD, Principal Investigator — UNC at Chapel Hill
Locations (1):
- Center for Infectious Disease Research in Zambia, Lusaka, Zambia

REFERENCES:
- [Derived] Mutale W, Ayles H, Lewis J, Bosompraph S, Chilengi R, Tembo MM, Sharp A, Chintu N, Stringer J. Protocol-driven primary care and community linkage to reduce all-cause mortality in rural Zambia: a stepped-wedge cluster randomized trial. Front Public Health. 2023 Aug 31;11:1214066. doi: 10.3389/fpubh.2023.1214066. eCollection 2023. PMID 37727608
- [Derived] Mutale W, Cleary S, Olivier J, Chilengi R, Gilson L. Implementing large-scale health system strengthening interventions: experience from the better health outcomes through mentoring and assessments (BHOMA) project in Zambia. BMC Health Serv Res. 2018 Oct 19;18(1):795. doi: 10.1186/s12913-018-3619-3. PMID 30340583
- [Derived] Mwanza M, Zulu J, Topp SM, Musonda P, Mutale W, Chilengi R. Use of Lot quality assurance sampling surveys to evaluate community health worker performance in rural Zambia: a case of Luangwa district. BMC Health Serv Res. 2017 Apr 17;17(1):279. doi: 10.1186/s12913-017-2229-9. PMID 28416009
- [Derived] Yan LD, Chirwa C, Chi BH, Bosomprah S, Sindano N, Mwanza M, Musatwe D, Mulenga M, Chilengi R. Hypertension management in rural primary care facilities in Zambia: a mixed methods study. BMC Health Serv Res. 2017 Feb 3;17(1):111. doi: 10.1186/s12913-017-2063-0. PMID 28158981
- [Derived] Mutale W, Stringer J, Chintu N, Chilengi R, Mwanamwenge MT, Kasese N, Balabanova D, Spicer N, Lewis J, Ayles H. Application of balanced scorecard in the evaluation of a complex health system intervention: 12 months post intervention findings from the BHOMA intervention: a cluster randomised trial in Zambia. PLoS One. 2014 Apr 21;9(4):e93977. doi: 10.1371/journal.pone.0093977. eCollection 2014. PMID 24751780